CLINICAL TRIAL: NCT03073109
Title: PATIENT-REPORTED OUTCOMES IN RHEUMATOID ARTHRITIS PATIENTS TREATED WITH TOFACITINIB OR BIOLOGICAL DISEASE-MODIFYING ANTIRHEUMATIC DRUGS (DMARDS) IN REAL LIFE CONDITIONS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921284
Record Dates: First submitted 2017-01-03; First posted 2017-03-08 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is aimed to describe the outcomes related to physical activity, activity of disease, quality of life, work productivity and safety in Latin-American patients with Rheumatoid Arthritis (RA) treated with tofacitinib or biological DMARDs after failure to respond to conventional DMARDs in real-life conditions. This will be a non-interventional, hybrid study (prospective and retrospective data collection) comparing tofacitinib to biologic DMARD treatments in patients with RA after failure of conventional DMARDs. The population will be composed by adult patients over 18 years of age diagnosed with RA and who have been prescribed tofacitinib or any biological DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age at the time of recruitment
* Patient diagnosed with moderate to severe RA ≥ 6 months before enrollment
* Patients who have had an inadequate response to the continuous use of methotrexate or combination of conventional DMARDs for at least 12 weeks before the study without dose change within the last 8 weeks before enrollment in the study
* Patients with no biological DMARDs use in patient history.
* Patients prescribed with tofacitinib or biological DMARDs in the last two weeks at doses established in ACR guidelines published in 2015 and following medical criteria.
* Acceptance for patients to participate in the study and signing of the informed consent.

Exclusion Criteria:

* Patients who do not have the ability to answer the questionnaires by themselves or who have any kind of mental disorder that may affect their answers.
* Patients diagnosed with autoimmune rheumatic diseases other than RA and Sjogren's syndrome.
* Patients treated with biological DMARDs in monotherapy.
* Participation in other studies involving investigational drug(s) (Phases 1-4) within 4 weeks or 5 half-lives (whichever is longer) after discontinuation of the investigational compound before the current study begins and/or during study participation.
* Patients with any current malignancy or a history of malignancy, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* Patients with lymphoproliferative disorders (e.g., Epstein Barr Virus (EBV) related lymphoproliferative disorder), a history of lymphoma, leukemia, or signs and symptoms suggestive of current lymphatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients ≥ 18 years of age diagnosed with RA and who failed to respond to conventional DMARDs, and have been prescribed tofacitinib or any biological DMARDs
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Colombia (10):
  - Artmedica, Medellín, Antioquia
  - Fundacion Instituto de Reumatologia Fernando Chalem, Bogota, Cundinamarca
  - IDEARG, Bogota, Cundinamarca
  - Clinica de Occidente, Cali, Valle del Cauca Department
  - Centro Integral de Reumatología del Caribe Circaribe S.A, Barranquilla
  - Clinicos IPS, Bogotá
  - Centro de Investigacion en Reumatologia y Especialidades Medicas S.A.S, CIREEM, Bogotá
  - SERVIMED, Bucaramanga
  - Fundacion Valle del Lili, Cali
  - REUMALAB, Medellín
- Peru (3):
  - Clínica San Judas Tadeo, Lima, SAN Miguel
  - Centro Medico CEEN, Arequipa
  - Clinica Jockey Salud, Lima

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Reyes JM, Gutierrez MV, Madariaga H, Otero W, Guzman R, Izquierdo J, Abello M, Velez P, Castillo D, Ponce de Leon D, Lukic T, Amador L. Patient-reported outcomes in RA patients treated with tofacitinib or bDMARDs in real-life conditions in two Latin American countries. Reumatol Clin (Engl Ed). 2023 Jun-Jul;19(6):319-327. doi: 10.1016/j.reumae.2023.02.006. PMID 37286268
- [Derived] Gutierrez-Ardila MV, Reyes J, Madariaga H, Otero W, Guzman R, Izquierdo J, Abello M, Velez P, Castillo D, Ponce de Leon D, Lukic T, Amador L. Work productivity in rheumatoid arthritis patients from two Latin American countries treated with tofacitinib or biological DMARDs. Expert Rev Pharmacoecon Outcomes Res. 2022 Jul;22(5):787-794. doi: 10.1080/14737167.2022.2047935. Epub 2022 Mar 16. PMID 35249439
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included participants from two Latin American countries (Colombia and Peru) from 15 March 2017 to 16 September 2019.
Pre-assignment Details: This was a non-interventional, hybrid study (prospective and retrospective data collection).
Groups:
- Tofacitinib: Participants with rheumatoid arthritis (RA) treated with tofacitinib after failure of conventional disease-modifying anti-rheumatic drugs (DMARDs) were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months.
- Biologics: Participants with RA treated with biological DMARDs after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months.
Period: Overall Study
Arm/Group | Tofacitinib | Biologics
Started | 100 | 70
Completed | 90 | 68
Not Completed | 10 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Other | 2 | 0
Not completed — Lost to Follow-up | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Tofacitinib: Participants with RA treated with tofacitinib after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib | Biologics | Total
Number analyzed (Participants) | 100 | 70 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (14.4) | 51.3 (12.6) | 53.5 (13.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 15 | 4 | 19
  Female | 85 | 65 | 150
  Unknown | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100 | 69 | 169
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latin American | 100 | 69 | 169
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Routine Assessment of Patient Index Data 3 (RAPID3) Score at Month 6
Description: Disease activity was assessed using RAPID3, which was based on participant-reported multi-dimensional health assessment questionnaire (MDHAQ). RAPID3 included 3 core data set measures of physical function, pain, and patient global estimate. Physical function=mean of scores from 10 individual questions on activities of daily living (each question scored from '0'=no difficulty to '3'=much difficulty), scores were transformed to give a total score=0 to 10, higher scores=greater difficulty. Pain and global estimate of health measured on Likert scale from '0'=no pain/feeling very well to '10'=pain as bad as it could be/ feeling very poorly, higher scores=greater difficulty/ worsening of condition. RAPID3 composite score: mean of physical function, pain, and global assessment scores, ranging from 0 to 10, higher values=greater disease activity. Data has been provided in terms of adjusted (consider impact of co-variables) and unadjusted mean (does not consider co-variables impact).
Time Frame: Baseline, Month 6
Population: Analysis was performed on all participants included in the study. Here, 'Number analyzed' = participants evaluable for this outcome measure (OM) at specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tofacitinib: Participants with RA treated with tofacitinib after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were treatment interruption, access limitation, previous methotrexate and complementary access.
- Biologics: Participants with RA treated with biological DMARDs after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were treatment interruption, access limitation, previous methotrexate and complementary access.
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 100 | 70
units on a scale
  Baseline - adjusted mean | 7.12 (0.39) | 5.95 (0.31)
  Baseline - unadjusted mean | 5.88 (0.22) | 5.94 (0.22)
  Change at Month 6 - adjusted mean: number analyzed (Participants) | 90 | 68
  Change at Month 6 - adjusted mean | -0.20 (0.70) | -0.32 (0.72)
  Change at Month 6 - unadjusted mean: number analyzed (Participants) | 90 | 68
  Change at Month 6 - unadjusted mean | -2.71 (0.26) | -3.28 (0.30)

2. Secondary Outcome: Adapted Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Month 6
Description: Functional status of participants was assessed using adapted HAQ-DI. Adapted HAQ-DI is a participant-reported questionnaire for the assessment of ability to perform tasks in 8 categories of daily living activities due to rheumatoid arthritis: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point Likert scale from 0 to 3, where 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by total number of domains answered. Total possible score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning. Data has been provided in terms of adjusted (consider impact of co-variables) and unadjusted mean (does not consider co-variables impact).
Time Frame: Month 6
Population: Analysis was performed on participants included in the study who were evaluable for adapted HAQ-DI at month 6. Hence, 'Overall number of participants analyzed' = Participants who had data available for this OM.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tofacitinib: Participants with RA treated with tofacitinib after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were time to supply, access limitation, methotrexate concomitant, chloro-quine concomitant and participant access.
- Biologics: Participants with RA treated with biological DMARDs after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were sensitive joints, leflunomide concomitant, chloro-quine concomitant and public access.
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 90 | 68
units on a scale
  Adjusted mean | 0.93 (0.13) | 0.77 (0.10)
  Unadjusted mean | 0.96 (0.08) | 0.78 (0.08)

3. Secondary Outcome: Change From Baseline in Adapted Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Month 6
Description: Functional status of participants was assessed using adapted HAQ-DI. Adapted HAQ-DI is a participant-reported questionnaire for the assessment of ability to perform tasks in 8 categories of daily living activities due to rheumatoid arthritis: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point Likert scale from 0 to 3, where 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by total number of domains answered. Total possible score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning. Data has been provided in terms of adjusted (consider impact of co-variable) and unadjusted mean (does not consider co-variable impact).
Time Frame: Baseline, Month 6
Population: Analysis was performed on all participants included in the study. Here, 'Number analyzed' = participants evaluable for this OM at specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tofacitinib: Participants with RA treated with tofacitinib after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variable considered for adjusted mean was access limitation.
- Biologics: Participants with RA treated with biological DMARDs after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variable considered for adjusted mean was access limitation.
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 100 | 70
units on a scale
  Baseline - adjusted mean | 1.63 (0.13) | 1.50 (0.10)
  Baseline - unadjusted mean | 1.62 (0.08) | 1.46 (0.08)
  Change at Month 6 - adjusted mean: number analyzed (Participants) | 90 | 68
  Change at Month 6 - adjusted mean | -0.56 (0.07) | -0.50 (0.08)
  Change at Month 6 - unadjusted mean: number analyzed (Participants) | 90 | 68
  Change at Month 6 - unadjusted mean | -0.66 (0.07) | -0.68 (0.08)

4. Secondary Outcome: European Quality of Life- 5 Dimension-3 Levels (EQ-5D-3L) Index Score at Month 6
Description: EQ-5D-3L is a standardized, participant-administered measure of self-reported health outcomes. It consists of two parts: EQ-5D index score (Part I) and the EQ-VAS (Part II). For Part I, i.e. EQ-5D-3L index score, participants rated their current health state on 5 single-item dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with each dimension having three levels of measure: 1= no problems, 2= some problems and 3= extreme problems. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score was transformed and results in a total index score range of 0 to 1.00; higher scores indicating a better health state. Data has been provided in terms of adjusted (consider impact of co-variables) and unadjusted mean (does not consider co-variables impact).
Time Frame: Month 6
Population: Analysis was performed on participants included in the study. Hence, 'Overall number of participants analyzed' = only those participants who had data available for this OM.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tofacitinib: Participants with RA treated with tofacitinib after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were interruption of treatment and time to supply.
- Biologics: Participants with RA treated with biological DMARDs after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variable considered for adjusted mean was public access.
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 90 | 68
units on a scale
  Adjusted mean | 0.54 (0.05) | 0.67 (0.04)
  Unadjusted mean | 0.63 (0.03) | 0.65 (0.04)

5. Secondary Outcome: Change From Baseline in European Quality of Life- 5 Dimension-3 Levels (EQ-5D-3L) Index Score at Month 6
Description: EQ-5D-3L is a standardized, participant-administered measure of self-reported health outcomes. It consists of two parts: EQ-5D index score (Part I) and the EQ-VAS (Part II). For Part I, i.e. EQ-5D-3L index score, participants rated their current health state on 5 single-item dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with each dimension having three levels of function:. 1=no problems, 2=some problems and 3=extreme problems. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score was transformed and results in a total index score range of 0 to 1.00; higher scores indicating a better health state. Data has been provided in terms of adjusted (consider impact of co-variables) and unadjusted mean (does not consider co-variables impact).
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tofacitinib: Participants with RA treated with tofacitinib after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were access limitation and interruption of treatment.
- Biologics: Participants with RA treated with biological DMARDs after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were access limitation and interruption of treatment.
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 100 | 70
units on a scale
  Baseline - adjusted mean | 0.19 (0.05) | 0.23 (0.04)
  Baseline - unadjusted mean | 0.30 (0.03) | 0.22 (0.04)
  Change at Month 6 - adjusted mean: number analyzed (Participants) | 90 | 68
  Change at Month 6 - adjusted mean | 0.23 (0.06) | 0.29 (0.06)
  Change at Month 6 - unadjusted mean: number analyzed (Participants) | 90 | 68
  Change at Month 6 - unadjusted mean | 0.35 (0.04) | 0.43 (0.05)

6. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire for Rheumatoid Arthritis (WPAI:RA) Scores at Month 6
Description: WPAI-RA: 6-questions participant rated questionnaire that measures effect of participant's RA on general health and symptom severity on work productivity and regular activities. Consisted of 6 questions, a binary question on current employment, 3 questions on hours of work and work-loss, and 2 questions based on 0-10 point scale to judge how RA affected productivity at work and outside of work (0 = no effect on work and 10 = completely prevented from working). It yielded four sub-scores: percent work time missed due to health (absenteeism), percent impairment while working (presenteeism), percent overall work impairment due to health (work productivity loss) and percent activity impairment due to health (daily activity impairment/loss). Sub-scores were expressed as an impairment percentage range from 0 to 100, where 0 = no impairment, 100 = completely impaired, higher scores=greater impairment and less productivity. Data has been provided in terms of adjusted and unadjusted mean.
Time Frame: Month 6
Population: Analysis was performed on participants included in the study. Here, 'Overall number of participants analyzed' = only those participants who had data available for this OM. 'Number analyzed' = participants evaluable for this OM at specified categories.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tofacitinib: Participants with RA treated with tofacitinib after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were participant access, years since diagnosis, age, chloroquine concomitant, interruption of treatment, time to supply, access limitation, neutrophils, start treatment, methotrexate concomitant and chloroquine concomitant.
- Biologics: Participants with RA treated with biological DMARDs after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were access limitation, years since diagnosis, leflunomide, chloroquine, chloroquine concomitant and public access.
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 90 | 68
units on a scale
  Absenteeism: adjusted mean: number analyzed (Participants) | 23 | 22
  Absenteeism: adjusted mean | 12.3 (8.83) | 10.8 (6.74)
  Absenteeism: unadjusted mean: number analyzed (Participants) | 23 | 22
  Absenteeism: unadjusted mean | 8.78 (6.95) | 10.8 (6.74)
  Presenteeism: adjusted mean: number analyzed (Participants) | 24 | 21
  Presenteeism: adjusted mean | 32.10 (8.82) | 27.7 (6.33)
  Presenteeism: unadjusted mean: number analyzed (Participants) | 24 | 21
  Presenteeism: unadjusted mean | 23.30 (5.76) | 27.7 (6.33)
  Productivity loss: adjusted mean: number analyzed (Participants) | 23 | 21
  Productivity loss: adjusted mean | 37.8 (10.25) | 26.9 (6.67)
  Productivity loss: unadjusted mean: number analyzed (Participants) | 23 | 21
  Productivity loss: unadjusted mean | 29.3 (6.67) | 26.9 (6.67)
  Activity loss: adjusted mean | 42.7 (4.34) | 31.0 (4.79)
  Activity loss: unadjusted mean | 35.7 (2.75) | 27.1 (3.01)

7. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire for Rheumatoid Arthritis (WPAI:RA) Scores at Month 6
Description: WPAI-RA: 6-questions participant rated questionnaire that measures effect of participant's RA on general health and symptom severity on work productivity and regular activities. Consisted of 6 questions, a binary question on current employment, 3 questions on hours of work and work-loss, and 2 questions based on 0-10 point scale to judge how RA affected productivity at work and outside of work (0 = no effect on work and 10 = completely prevented from working). It yielded four sub-scores: percent work time missed due to health (absenteeism), percent impairment while working (presenteeism), percent overall work impairment due to health (work productivity loss) and percent activity impairment due to health (daily activity impairment/loss). Sub-scores were expressed as an impairment percentage range from 0 to 100, where 0 = no impairment, 100 = completely impaired, higher numbers=greater impairment and less productivity. Data has been provided in terms of adjusted and unadjusted mean.
Time Frame: Baseline, Month 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 99 | 70
units on a scale
  Absenteeism: Baseline - adjusted: number analyzed (Participants) | 27 | 28
  Absenteeism: Baseline - adjusted | 35.20 (8.59) | 36.10 (5.98)
  Absenteeism: Baseline - unadjusted: number analyzed (Participants) | 27 | 28
  Absenteeism: Baseline - unadjusted | 31.49 (6.41) | 36.10 (5.98)
  Absenteeism: Change at Month 6- adjusted: number analyzed (Participants) | 22 | 22
  Absenteeism: Change at Month 6- adjusted | -18.4 (7.74) | -19.4 (7.99)
  Absenteeism: Change at Month 6- unadjusted: number analyzed (Participants) | 22 | 22
  Absenteeism: Change at Month 6- unadjusted | -22.4 (7.02) | -24.2 (7.02)
  Presenteeism: Baseline - adjusted: number analyzed (Participants) | 28 | 26
  Presenteeism: Baseline - adjusted | 66.7 (8.35) | 59.2 (5.82)
  Presenteeism: Baseline - unadjusted: number analyzed (Participants) | 28 | 26
  Presenteeism: Baseline - unadjusted | 56.4 (5.33) | 59.2 (5.82)
  Presenteeism: Change at Month 6- adjusted: number analyzed (Participants) | 23 | 21
  Presenteeism: Change at Month 6- adjusted | -34.8 (5.89) | -34.8 (6.16)
  Presenteeism: Change at Month 6- unadjusted: number analyzed (Participants) | 23 | 21
  Presenteeism: Change at Month 6- unadjusted | -34.8 (5.89) | -34.8 (6.16)
  Productivity loss: Baseline - adjusted: number analyzed (Participants) | 27 | 26
  Productivity loss: Baseline - adjusted | 71.1 (9.69) | 65.1 (5.98)
  Productivity loss: Baseline - unadjusted: number analyzed (Participants) | 27 | 26
  Productivity loss: Baseline - unadjusted | 62.8 (6.15) | 65.1 (5.98)
  Productivity loss: Change at Month 6- adjusted: number analyzed (Participants) | 23 | 21
  Productivity loss: Change at Month 6- adjusted | -11.0 (16.5) | -15.9 (15.2)
  Productivity loss: Change at Month 6- unadjusted: number analyzed (Participants) | 23 | 21
  Productivity loss: Change at Month 6- unadjusted | -36.9 (6.47) | -39.2 (6.79)
  Activity loss: Baseline - adjusted | 78.0 (4.43) | 70.1 (4.79)
  Activity loss: Baseline - unadjusted | 67.1 (2.64) | 66.2 (3.01)
  Activity loss: Change at Month 6- adjusted: number analyzed (Participants) | 90 | 68
  Activity loss: Change at Month 6- adjusted | -43.80 (11.00) | -49.90 (13.30)
  Activity loss: Change at Month 6- unadjusted: number analyzed (Participants) | 90 | 68
  Activity loss: Change at Month 6- unadjusted | -32.80 (3.18) | -38.40 (3.66)

8. Secondary Outcome: Disease Activity Score Based on 28-joints Count (DAS28) at Month 6
Description: DAS28 calculated from the number of swollen joints and painful joints using the 28 joints count, erythrocyte sedimentation rate (ESR) (measured in millimeters per hour [mm/hour]) and patient's global assessment of disease activity according to 100-millimeter (mm) Visual Analog Scale (VAS) (scores ranging 0 [very well] to 100 mm [extremely bad], higher scores=worsening of condition). DAS28-ESR scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. DAS28 scores ranged from 0 to 10; higher scores indicated greater affectation due to disease activity. Data has been provided in terms of adjusted and unadjusted mean.
Time Frame: Month 6
Population: Analysis was performed on participants included in the study. Here, 'Overall number of participants analyzed' = only those participants who had data available for this OM.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tofacitinib: Participants with RA treated with tofacitinib after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were interruption of treatment, time to supply, access limitation, lymphocytes, neutrophils, swollen joints and corticoids concomitant.
- Biologics: Participants with RA treated with biological DMARDs after failure of conventional DMARDs were assessed for patient-reported outcomes in this study. Data for these participants was collected for approximately 2.5 years (from 15 March 2017 to 16 September 2019) and participants were followed up to 6 months. The co-variables considered for adjusted mean were time to supply, sensitive joints and public access.
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 86 | 61
units on a scale
  Adjusted Mean | 3.02 (0.24) | 2.61 (0.12)
  Unadjusted Mean | 3.10 (0.13) | 2.88 (0.43)

9. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-joints Count (DAS28) at Month 6
Description: as for outcome 8
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 100 | 70
units on a scale
  Baseline - adjusted mean | 5.59 (0.22) | 5.21 (0.11)
  Baseline - unadjusted mean | 5.21 (0.12) | 5.88 (0.40)
  Change at Month 6 - adjusted mean: number analyzed (Participants) | 86 | 61
  Change at Month 6 - adjusted mean | -3.86 (0.59) | -4.23 (0.61)
  Change at Month 6 - unadjusted mean: number analyzed (Participants) | 86 | 61
  Change at Month 6 - unadjusted mean | -2.13 (0.35) | -3.03 (0.42)

10. Secondary Outcome: Number of Participants With Serious Adverse Event (SAE) and Non-serious Adverse Events (AEs)
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs included both serious and non-serious adverse event. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Month 6
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 100 | 70
Participants
  Participants with SAE | 1 | 0
  Participants with Non-Serious AE | 20 | 16

11. Secondary Outcome: Number of Participants With Serious Infections
Description: Serious infection defined as any infection that requires hospitalization.
Time Frame: Baseline up to Month 6
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 100 | 70
Participants | 1 | 0

12. Secondary Outcome: Number of Participants Who Withdrew From Study Due to Adverse Events And Due to All Causes
Description: Here, number of participants who withdrew from study due to AEs and due to all causes (withdrawals due to AEs, lost to follow up and unspecified reasons) have been described.
Time Frame: Baseline up to Month 6
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Biologics
Number analyzed (Participants) | 100 | 70
Participants
  Due to AEs | 0 | 1
  Due to All causes | 10 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to Month 6
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Tofacitinib | Biologics
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/70
Serious Adverse Events (participants affected / at risk) | 1/100 | 0/70
Other Adverse Events (participants affected / at risk) | 20/100 | 16/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib (N=100) | Biologics (N=70)
Appendicitis (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib (N=100) | Biologics (N=70)
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Purpura (Blood and lymphatic system disorders) | 1 | 0
Oligomenorrhea (Endocrine disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 3
Malaise (General disorders) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Spinal pain (Nervous system disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 2
Vulvovaginitis (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pharyngitis bacterial (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngotonsillitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
DAS 28 data for month 3 was not collected and analyzed since data was planned to be collected depending on the availability of medical records as specified in analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT03073109/Prot_SAP_000.pdf